CLINICAL TRIAL: NCT04252053
Title: The Effects of Pilates-Based Core Stabilization Training on Isokinetic Knee Strength and Postural Sway in People With Multiple Sclerosis
Brief Title: The Effects of Pilates-Based Core Stabilization Training in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Feray Güngör, Physiotherapist, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59491012-604.01.02-
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Pilates; Core stability; Isokinetic strength; Postural sway
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Pilates-Based Core Stability Training Group (Experimental): In order to detect the effects of pilates-based core stabilization training (PBCST) on isokinetic knee strength and postural sways, individuals with MS will receive pilates-based core stabilization training for 8 weeks and 2 days a week. One educational session will perform to teach basic principles of pilates based training. Individuals in this group will receive treatment at the clinic by physiotherapist supervision. All sessions will be individualized (not group training).
  Interventions: Other: Pilates Based Core Stabilization Training
- Home exercise group (Active Comparator): The home exercise group will perform the same PBCST exercises at home during the same period (8 weeks, 2 days a week) as the brochures prepared for them. Individuals in this group will receive one educational session which includes basic principles of pilates and one session which includes two-week exercise program. Participants will be invited to the clinic every two weeks to ensure the progression of the exercises and the exercise program will be updated.
  Interventions: Other: Home based exercise

INTERVENTIONS:
Other: Pilates Based Core Stabilization Training — Pilates-based core stabilization training (PBCST) is a controlled form of exercise provided improvement in stabilization of abdominal and back muscles.
  Arms: Supervised Pilates-Based Core Stability Training Group
Other: Home based exercise — Home exercises which include pilates based core stabilization training will be structured for the people with MS according to their physical condition and will perform at home by them.
  Arms: Home exercise group

SUMMARY:
Multiple Sclerosis (MS) is a chronic, autoimmune and neurodegenerative disease characterized by inflammation and progressive demyelination of the central nervous system. It is characterized by muscle weakness, balance and coordination disorder, which is more common in the lower extremities and trunk muscles. Over time, these symptoms decrease the individual's level of physical activity, mobility and quality of life, leading to further deterioration of the disorder. One of the most important problems that cause these problems in individuals with MS is reduced core stabilization. Decrease in core stabilization affects the quality of limb movements as well as trunk stability when considering the kinetic chain in the body. Pilates-based core stabilization training (PBCST) are a controlled exercise form used to improve the stabilization of trunk muscles. There are no studies on the effect of this training on lower extremity isokinetic muscle strength in individuals with MS. The aim of this study is to determine the effect of PBCST on lower extremity muscle strength, postural sway and kinetic chain in individuals with MS.

DETAILED DESCRIPTION:
The study was planned as randomized controlled. Individuals included in the study wiil randomly allocate to the group receiving the supervised PBCST and the home exercise group. While the supervised exercise group receives PBCST for 2 days and 8 weeks in the clinic, the home exercise group will perform the same exercises at home for the same time as the brochures prepared for them. The exercise program will show progression at 2-week intervals. A session will be held for both groups to teach the basic principles of pilates and will not be counted in the 8-week program. At the beginning and end of treatment, individuals will be evaluated for isokinetic muscle strength, balance and postural sway, fatigue level, quality of life and functional capacity parameters. PBCST is thought to reduce postural sways and increase lower extremity muscle strength by increasing core stability with the effect of kinetic chain and increased stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MS according to McDonald's criteria
* Disability level less than 6 according to EDSS (Expanded Disability Status Scale) score
* No attacks during the last 3 months
* Being an ambulatory
* Volunteering to participate in the study

Exclusion Criteria:

* Having orthopedic, neurological, psychological, etc. diseases that accompany MS and may affect treatment outcomes
* Doing regular sports
* Being involved in another physiotherapy and rehabilitation program related to MS

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Isokinetic strength | 8 weeks
  Concentric isokinetic muscle strength of the knee flexor and extensor muscles will be evaluated at angular velocities of 30,60 and 90°/s.
Postural sways | 8 weeks
  Postural sways will be evaluated with biodex balance system in different condition such as open eyes on firm and foam surface, closed eyes on firm and foam surface, tandem stance on firm and foam surface,

SECONDARY OUTCOMES:
Core strength | 8 weeks
  Core strength will be evaluated within the scope of core assessment. Curl-Up and Modified Push-Up test will be used for the evaluation of core strength.
Core endurance | 8 weeks
  Core endurance will be evaluated within the scope of core assessment. Trunk Flexor Endurance Test, Trunk Extensor Endurance Test, Trunk Lateral Endurance Test and Plank Test will be used in the evaluation of core endurance.
Balance | 8 weeks
  Berg Balance Scale (BBS) will be used to evaluate balance. BBS is a test developed for functional evaluation of balance in adults. BBS consists of 14 general equilibrium activities that change the orientation of the body center of gravity relative to the support surface and the ability to maintain the static position during the reduction of the support surface. The highest score is 56. The decrease in the score indicates poorer balance.
Mobility | 8 weeks
  Two-minute walk test (2-MWT) will be used to evaluate the mobility of the people with MS. 2-MWT is a measure of self-paced walking ability and functional capacity.
Fatigue | 8 weeks
  Fatigue Severity Scale (FSS) will be used to evaluate fatigue levels. This scale evaluates the severity of fatigue with 9 questions. Each question scores between 1 (I do not agree) and 7 (fully agree). The FSS score is the average value of nine sections. A high score indicates increased fatigue severity.
Quality of life | 8 weeks
  Multiple Sclerosis Quality of Life -54 (MSQOL-54) will be used to evaluate the effectiveness of the treatment on quality of life. The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument.
Fall risk | 8 weeks
  Timed Up and Go (TUG) will be used. TUG is a test used to determine fall risk and measure the progress of balance, sit to stand and walking.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)